CLINICAL TRIAL: NCT00316823
Title: Gene Expression Analysis in Thyroid Nodule FNA Samples
Brief Title: Genetic Analysis in Diagnosing Thyroid Cancer in Patients With Thyroid Nodules
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Diagnostic
Other Study IDs: CDR0000456480; UCSF-H28355-27029-01; UCSF-05205
Record Dates: First submitted 2006-04-19; First posted 2006-04-21 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2008-12

CONDITIONS: Head and Neck Cancer
Keywords: thyroid cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Thyroid Neoplasms | interventions — Gene Expression Profiling; Polymerase Chain Reaction; Reverse Transcriptase Polymerase Chain Reaction; Immunohistochemistry; Biopsy, Needle

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: polymerase chain reaction
Genetic: reverse transcriptase-polymerase chain reaction
Other: diagnostic laboratory biomarker analysis
Other: immunohistochemistry staining method
Procedure: needle biopsy

SUMMARY:
RATIONALE: Finding genetic markers for thyroid cancer in a biopsy specimen may help doctors diagnose thyroid cancer.

PURPOSE: This clinical trial is studying how well genetic analysis works in diagnosing thyroid cancer in patients with thyroid nodules.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the diagnostic accuracy of biomarkers and mRNA expression analysis using fine-needle aspiration (FNA) biopsy samples from patients with thyroid nodules.
* Correlate the level of gene expression with the aggressiveness of differentiated thyroid cancer in FNA biopsy samples.

OUTLINE: Patients undergo fine-needle aspiration (FNA) biopsy as part of routine care. Additional thyroid tissue is collected during the biopsy for gene expression analysis. Patients who have already had a biopsy undergo FNA biopsy during thyroidectomy.

Tissue samples will be examined for gene expression by reverse transcriptase-polymerase chain reaction (PCR), real-time quantitative PCR, and immunohistochemistry.

PROJECTED ACCRUAL: A total of 400 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of a thyroid nodule that requires fine-needle aspiration biopsy or thyroidectomy to exclude a diagnosis of thyroid cancer

PATIENT CHARACTERISTICS:

* Platelet count ≥ 70,000/mm^3
* PT (INR) ≤ 14.5
* PTT ≤ 35.2
* Not pregnant

PRIOR CONCURRENT THERAPY:

* No aspirin or nonsteroidal anti-inflammatory drugs (NSAIDs) 7 days before sample procurement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2005-07; Primary Completion 2009-12

PRIMARY OUTCOMES:
Diagnostic accuracy of biomarkers by mRNA expression analysis
Correlate levels of gene expression with the aggressiveness of differentiated thyroid cancer in FNA biopsy samples

CONTACTS AND LOCATIONS:
Overall Officials: Electron Kebebew, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States